CLINICAL TRIAL: NCT03575234
Title: Phase I Neo-Adjuvant Nivolumab + IRX-2 Followed by Surgery for Resectable Oral Cavity Cancer or HPV-Associated Oropharynx Cancer
Brief Title: Nivolumab & IRX-2 With Surgery for Resectable Stage III-IVA Oral Cavity Cancer or HPV-Positive Oropharyngeal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: funding and drug were withdrawn
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Brooklyn ImmunoTherapeutics, LLC (Industry)
Responsible Party: Principal Investigator, Mihir Patel, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00102105; NCI-2018-00411 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4300-18 (Other: Emory University Hospital/Winship Cancer Institute)
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Human Papillomavirus Positive Oropharyngeal Squamous Cell Carcinoma; Stage II Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage IVA Oral Cavity Squamous Cell Carcinoma AJCC v6 and v7; Stage III Oropharyngeal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cyclophosphamide; IRX 2; Nivolumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, cyclophosphamide, IRX-2, surgery) (Experimental): Participants receive nivolumab IV over 60 minutes on days 1 and 15, cyclophosphamide IV on day 1, and IRX-2 SC over 10 consecutive days between days 4-21 in the absence of disease progression or unacceptable toxicity. Beginning days 25-30, participants undergo surgery.
  Interventions: Drug: Cyclophosphamide; Biological: IRX-2; Biological: Nivolumab; Procedure: Surgery

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: Cytophosphane; Cytoxan; Neosar; Revimmune
Biological: IRX-2 — Given SC
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; ONO-4538; Opdivo
Procedure: Surgery — Undergo surgery

SUMMARY:
This phase I trial studies the side effects of nivolumab and IRX-2 and how well they work in treating participants with stage III-IVA oral cavity cancer or human papillomavirus (HPV)-positive oropharyngeal cancer that can be removed by surgery. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread. IRX-2 may "turn on" the immune system and stimulate an immune response against tumor cells. Giving nivolumab and IRX-2 followed by surgery may work better at treating oral cavity and oropharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of combination immunotherapy, nivolumab + IRX-2, for HPV+ oropharyngeal squamous cell carcinoma (OPSCC) and HPV- oral cavity squamous cell carcinoma (OCSCC).

II. To assess the oncologic efficacy of neo-adjuvant immunotherapy using pathologic confirmation of response after surgical resection.

SECONDARY OBJECTIVES:

I. To correlate tumor microenvironment histopathology with pathologic findings, with progression free survival (PFS) and other outcome parameters in patients with resectable OPSCC and OCSCC after the above treatments.

II. To evaluate swallowing function before and after surgery and risk-adjusted adjuvant therapy.

III. To evaluate quality of life (QOL), swallowing perception and performance, voice outcomes, and head and neck symptoms.

OUTLINE: Participants receive nivolumab intravenously (IV) over 60 minutes on days 1 and 15, cyclophosphamide IV on day 1, and IRX-2 subcutaneously (SC) over 10 consecutive days between days 4-21 in the absence of disease progression or unacceptable toxicity. Beginning days 25-30, participants undergo surgery.

After completion of study treatment, patients are followed up at 3 months, every 3 months for 2 years, then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Pathologically confirmed (histology or cytology), p16-negative (by immunohistochemistry [IHC]) stage II, III, or IVA squamous cell cancer of the oral cavity (excluding lip)
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Disease is surgically resectable with curative intent
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Hemoglobin > 9 g/dL
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Lymphocyte count > 500/µL
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Neutrophil count > 1500/µL
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Platelet count > 100,000/µL
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Serum albumin > 3.0 g/dL
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Aspartate aminotransferase (AST/serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT/ serum glutamate pyruvate transaminase [SGPT]) < 3 x the upper limits of normal (ULN)
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Alkaline phosphatase < 2 x ULN
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Prothrombin time (PT) and partial thromboplastin time (PTT) < 1.4 x ULN
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Calculated creatinine clearance > 50 mL/min
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Willing and able to give informed consent and adhere to protocol therapy
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Eastern Cooperative Oncology Group (ECOG) performance status < 2
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Female of childbearing potential (less than 12 months post-menopausal) or male with a partner of childbearing potential either agrees to be abstinent or uses a medically acceptable form of birth control during the study and for a period of 1 year
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Negative urine/serum pregnancy test (female participants only) at the time of screening and within 24 hours of study treatment, if applicable
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Stage 1 (T1/2 N1) squamous cell carcinoma of the oropharynx associated with HPV as determined by p16 protein expression using immunohistochemistry (IHC) performed by a Clinical Laboratory Improvement Amendments [CLIA] approved laboratory
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: No prior radiation above the clavicles
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Patients with a history of a curatively treated malignancy must be disease-free for at least two years prior to entry on study except for carcinoma in situ of cervix, melanoma in-situ (if fully resected), and/or non-melanomatous skin cancer
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Patients must not have evidence of extensive or "matted/fixed" pathologic adenopathy on preoperative imaging
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Hemoglobin > 9 g/dL
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Lymphocyte count > 500/µL
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Neutrophil count > 1500/µL
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Platelet count > 100,000/µL
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Serum albumin > 3.0 g/dL
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Aspartate aminotransferase (AST/ SGOT) and alanine aminotransferase (ALT/ SGPT) < 3 x the upper limits of normal (ULN)
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Alkaline phosphatase < 2 x ULN
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Prothrombin time (PT) and partial thromboplastin time (PTT) < 1.4 x ULN
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Calculated creatinine clearance > 50 mL/min
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Willing and able to give informed consent and adhere to protocol therapy
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: ECOG performance status < 2
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Female of childbearing potential (less than 12 months post-menopausal) or male with a partner of childbearing potential either agrees to be abstinent or uses a medically acceptable form of birth control during the study and for a period of 1 year
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Negative urine/serum pregnancy test (female participants only) at the time of screening and within 24 hours of study treatment, if applicable

Exclusion Criteria:

* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Prior surgery, radiation therapy, or chemotherapy other than biopsy or emergency procedure required for supportive care
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte associated protein 4 (anti-CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Prior treatment with cetuximab or epidermal growth factor receptor (EGFR) inhibitors in any treatment setting
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Any medical contraindications or previous therapy that would preclude treatment with either nivolumab, IRX-2, the surgery, reconstruction or adjuvant therapy required to treat the oral tumor appropriately
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Clinical status of either subject or tumor such that administration of 10 day neoadjuvant IRX-2 before surgery would be medically inappropriate
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Primary tumor of the oropharynx
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Tumor involvement of the following sites or any of these signs or symptoms likely to be associated with T4b cancer:

  * Involvement of pterygopalatine fossa, maxillary sinus, or facial skin
  * Gross extension of tumor to the skull base
  * Pterygoid plate erosion
  * Sphenoid bone or foramen ovale involvement
  * Direct extension to involve prevertebral fascia
  * Extension to superior nasopharynx or Eustachian tube
  * Direct extension into the neck with involvement of the deep neck musculature (neck node fixation)
  * Suspected invasion (encasement) of the common or internal carotid arteries; encasement will be assessed radiographically and will be defined as tumor surrounding the carotid artery 270 degrees or greater
  * Direct extension of neck disease to involve the external skin
  * Direct extension to mediastinal structures
  * Regional metastases to the supraclavicular neck (low level VB and IVB)
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Any investigational agent within the previous 30 days
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Daily administration of systemic immunosuppressive therapy or corticosteroids (except in physiological doses for hormone deficiency) during the previous 30 days
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Chronic anticoagulation, not including aspirin, but including heparins, warfarin, oral anticoagulation or other platelet function inhibitors
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Symptomatic cardiopulmonary disease (including congestive heart failure and hypertension), coronary artery disease, serious arrhythmia or chronic lung disease; patients with these conditions who are stable with relatively minor symptoms and who are appropriate candidates for surgical treatment of their tumor need not be excluded
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Myocardial infarction within the last 3 months
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Evidence of distant metastases (M1 disease) or other concurrent primary malignancy
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Known infection with hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Signs or symptoms of systemic infection (use of antibiotics to treat superficial infection or contamination of tumor shall not, by itself, be considered evidence of infection
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Stroke or other symptoms of cerebral vascular insufficiency within the last 3 months
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Allergy to ciprofloxacin (or other quinolones) and acetylsalicylic acid
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Previous diagnosis of invasive cancer from which the individual is NOT disease-free AND that has required treatment within the past 5 years, except for superficial skin, cervical cancer in-situ, well-differentiated thyroid or early stage prostate or bladder cancer (i.e., treatment with curative intent and long term disease-free expectations)
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: Prior axillary dissection
* ORAL CAVITY SQUAMOUS CELL CARCINOMA COHORT: History of pneumonitis or interstitial lung disease
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Prior surgery, radiation therapy, or chemotherapy other than biopsy or emergency procedure required for supportive care
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Any medical contraindications or previous therapy that would preclude treatment with either nivolumab or IRX-2 or the surgery, reconstruction or adjuvant therapy required to treat the oropharynx tumor appropriately
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Tumor of the oral cavity
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Tumor involvement of the following sites or any of these signs or symptoms likely to be associated with T4b cancer:

  * Involvement of pterygopalatine fossa, maxillary sinus
  * Gross extension of tumor to the skull base
  * Pterygoid plate erosion
  * Sphenoid bone or foramen ovale involvement
  * Direct extension to involve prevertebral fascia
  * Extension to superior nasopharynx or Eustachian tube
  * Direct extension into the neck with involvement of the deep neck musculature (neck node fixation)
  * Suspected invasion (encasement) of the common or internal carotid arteries; encasement will be assessed radiographically and will be defined as tumor surrounding the carotid artery 270 degrees or greater
  * Direct extension of neck disease to involve the external skin
  * Direct extension to mediastinal structures
  * Regional metastases to the supraclavicular neck (low level VB and IVB)
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Any investigational agent within the previous 30 days
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Daily administration of systemic immunosuppressive therapy or corticosteroids (except in physiological doses for hormone deficiency) during the previous 30 days
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Chronic anticoagulation, not including aspirin, but including heparins, warfarin, oral anticoagulation or other platelet function inhibitors
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Symptomatic cardiopulmonary disease (including congestive heart failure and hypertension), coronary artery disease, serious arrhythmia or chronic lung disease; patients with these conditions who are stable with relatively minor symptoms and who are appropriate candidates for surgical treatment of their tumor need not be excluded
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Myocardial infarction within the last 3 months
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Evidence of distant metastases (M1 disease) or other concurrent primary malignancy
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Known infection with hepatitis B, hepatitis C, or HIV
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Signs or symptoms of systemic bacterial infection (use of antibiotics to treat superficial infection or contamination of tumor shall not, by itself, be considered evidence of infection)
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Stroke or other symptoms of cerebral vascular insufficiency within the last 3 months
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Allergy to ciprofloxacin (or other quinolones), acetylsalicylic acid
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Previous diagnosis of invasive cancer from which the individual is NOT disease-free AND that has required treatment within the past 5 years, except for superficial skin, cervical cancer in-situ, well-differentiated thyroid or early stage prostate or bladder cancer (i.e., treatment with curative intent and long term disease-free expectations)
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: Prior axillary dissection
* HPV-ASSOCIATED OROPHARYNX SQUAMOUS CELL CARCINOMA COHORT: History of pneumonitis or interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) described using Common Terminology Criteria for Adverse Events 4.03 | Up to 4 years
  Non-hematologic toxicities will be evaluated via the ordinal Common Toxicity Criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level and patient will be explored and summarized.
Change in tumor size determined by central radiology review by radiologists blinded to the treatment regimen | Baseline up to 4 years
  Tumor changes will be determined by a comparison of the imaging studies (contrast-enhanced computed tomography [CECT] or magnetic resonance imaging [MRI]) obtained pre-treatment and just prior to surgery. Percent changes in tumor size will be determined by radiology at the site. If the change is not clear to the radiologist at the site, then the PI must be notified and two radiologists at Emory will be asked to independently review the scans and a decision will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Mihir Patel, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia